CLINICAL TRIAL: NCT02006433
Title: Treatment of Pain and Autonomic Dysreflexia in Spinal Cord Injury With Deep Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Jagid (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jonathan Jagid, Associate Professor of Neurological Surgery and Neurology, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20120429; W81XWH-12-1-0559 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2013-10-25; First posted 2013-12-10 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pain; Autonomic Dysreflexia
MeSH Terms: conditions — Pain; Autonomic Dysreflexia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Deep Brain Stimulation (Experimental): Deep brain stimulation (DBS) for the alleviation of chronic neuropathic pain in patients with spinal cord injury (SCI). The stimulation will be applied bilaterally or unilaterally in the midbrain periaqueductal/periventricular gray region (PAG/PVG).
  Extended participation in the study, which will last approximately 2 more years, precisely 104 weeks.The purpose of this extended portion of the study is to obtain long-term follow-up information on safety and efficacy, in subjects that have opted to receive continuing brain stimulation. Investigators label weeks in terms of original enrollment. Thus the surgery occurs in weeks 7 and 8 and the original study finishes in week 52, with the extension lasting from week 53 to week 156.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Local anesthesis, MRI and CT scan of the brain followed by implantation of the stimulation device
  Other Names: The Medtronic Models 3387 and 3389 DBS Leads neurostimulation system for deep brain stimulation.

SUMMARY:
The purpose of this research study is to determine if DBS is a feasible, safe and effective therapy for pain and autonomic dysreflexia after spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22-60 years of age
2. Level of injury at or above T12
3. Neuropathic pain at or below the level of injury, as determined based on pain in an area with neurological deficit and described as burning, shooting, electric, stinging etc.
4. The injury must have occurred at least 1 year prior to entering the study and participants must have experienced chronic pain for a minimum of six months.
5. The injury level must be at or above T12, and the disability must have a grade on the American Spinal Injury Association Impairment Scale (AIS) of ASIA-A, ASIA-B, ASIA-C or ASIA-D as determined by a qualified examiners.
6. Autonomic dysreflexia can be present, but is not a requirement. This is defined as a rise of systolic pressure by more than 30 mmHg during noxious skin stimulation or when the bladder or bowel is full, or apparently spontaneously over a period of minutes.
7. Pain (neuropathic) of moderate severity or greater is present, when the patient is taking medication, with a score of at least 4 on a numerical rating scale (range of 0 to 10).
8. Treatment with at least two of the following drug classes must have failed to give satisfactory pain relief within the last two years: anticonvulsants e.g., pregabalin, gabapentin); antidepressants (e.g., trazodone, amitriptyline); NSAIDS (e.g., ibuprofen). In addition, at least one of the following must have proved ineffective: exercise-based rehabilitation, massage therapy using a variety of methods, acupuncture using pressure, needles, heat, or electrical stimulation on specific points on the body and psychological interventions such as cognitive therapy.
9. The subject must be taking pain medication to maintain a stable level of medication from 4 weeks before surgery to 12 weeks after (the primary endpoint), except on the day of surgery.
10. Participants on medications for other conditions, such as diabetes, will be considered as candidates for this study. The dose will be monitored throughout the trial. (They will be excluded if the drug is being used to treat epilepsy, Parkinson's diseases, or other brain degenerative diseases.)
11. The subject must be willing to comply with the protocol including all scheduled visits.
12. Literate at 8th grade level or above.
13. Subject must provide a letter of clearance for the DBS surgery from primary care physician

Exclusion Criteria for Admission to study:

1. Unable to give informed consent
2. Prisoner or ward of the state
3. Pregnancy
4. Prior history of abusing nonprescribed drugs
5. Recent (one-year) history of alcohol abuse
6. ASIA motor exam unobtainable
7. History of cardiac arrhythmia
8. Renal disease, heart disease or uncontrolled hypertension (except due to autonomic dysreflexia), liver disease or hepatic cirrhosis
9. Active major medical or psychiatric illness
10. Significant post-traumatic encephalopathy from head trauma sustained at SCI
11. Languages without local expertise
12. Pain is only nociceptive, or due to muscle spasms

Exclusion Criteria for Treatment/Intervention procedure:

1. Coagulopathy requiring anticoagulation therapy
2. Thrombocytopenia or platelet dysfunction
3. Peripheral vascular disease
4. Comorbid neurological diseases or disorders, including a history of seizures
5. Active systemic infection or concurrent immunosuppressive therapy
6. Existing implantable cardiac pacemaker, defibrillator,or neurostimulator
7. Requiring short-wave or microwave diathermy treatment
8. Inability to cooperate
9. Any contraindication to MRI studies (All future MRIs, with the exception of brain MRIs, are excluded.)
10. Adverse reaction to stimulation (such as inability to stimulate at analgesic levels without causing clinical hypertension or hypotension) or allergy or hypersensitivity to any materials of the neurostimulation system
11. Depression, as defined by a Beck Depression Inventory (BDI-1a) score above 30.
12. Subjects with any clinically significant abnormality, not expected on the basis of age (age-related), that is seen in magnetic resonance imaging (MRI).

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2013-12; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in Pain as measured by Neuropathic Pain Symptom Inventory (NPSI) | Baseline, up to 52 weeks
  Neuropathic Pain Symptom Inventory (NPSI) is a 12 item questionnaire with each question scored form 0-10 with the highest score indicating greater pain
Change in Pain as measured by Multidimensional pain Inventory (MPI-SCI) | Baseline, up to 52 weeks
  Multidimensional pain Inventory (MPI-SCI) is a self-report questionnaire consisting of 50 items, each questioned scored from 0-6, with the higher score being the greatest impact of pain on an individuals daily life.
Change in Pain as measured by the Basic Pain Data Set | Baseline, up to 52 weeks
  The Basic Pain Data set is a 4 question assessing change in pain in the past week using 0-6 scale on each item with the higher score indicating greater pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan R Jagid, M.D., Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami Hospital, Miami, Florida
  - VA Medical Center, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT02006433/Prot_SAP_000.pdf